CLINICAL TRIAL: NCT04006756
Title: BrainFit: The Effect of Online Cognitive Training in Patients With Late Life Mood Disorders.
Brief Title: A Study on Better Cognitive Functioning Through Braintraining on the Internet
Acronym: BrainFit
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Amsterdam UMC, location VUmc (Other)
Responsible Party: Principal Investigator, Annemiek Dols, MD, PhD, Psychiatrist, Prinicipal Investigator, Amsterdam UMC, location VUmc
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NL58750.029.16
Record Dates: First submitted 2019-02-12; First posted 2019-07-05 (Actual); Last update posted 2021-12-01 (Actual); Status verified 2021-11

CONDITIONS: Depression; Late Life Mood Disorder; Impaired Cognition; Alteration in Mood; Alteration in Cognition
MeSH Terms: conditions — Depression; Cognition Disorders

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Online cognitive training 1 (Experimental): Eight-week, three times a week during 45 minutes cognitive training
  Interventions: Behavioral: Online cognitive training 1
- Online cognitive training 2 (Active Comparator): Eight-week, three times a week during 45 minutes cognitive activities
  Interventions: Behavioral: Online cognitive training 2

INTERVENTIONS:
Behavioral: Online cognitive training 1 — Eight-week online cognitive training program, three times a week for 45 minutes. The training contains several games that are designed to train cognitive functions.
  Arms: Online cognitive training 1
Behavioral: Online cognitive training 2 — Eight-week online active comparator program, three times a week for 45 minutes. The training contains several games.
  Arms: Online cognitive training 2

SUMMARY:
This study evaluates the efficacy of an eight-week online cognitive training program on feasability and on objective and subjective cognitive functions in patients with late life mood disorders (LLMD). In the feasability study two training groups will be compared. The primary aim is to investigate feasability, measured by compliance attendance and satisfaction of the participants. The secondary aim is to study the possible effects of the intervention on cognitive functions. Additionally, effects on mood symptoms, social functioning, sense of mastery and quality of lide will be studied.

DETAILED DESCRIPTION:
BACKGROUND OF THE STUDY Late life mood disorders (LLMD) include patients with unipolar depression and bipolar disorder, aged 50 years and over. Despite the fact that evidence-based pharmacological and psychotherapeutic interventions have proven effective, many patients with LLMD experience relapse or partial remission.

One of the reasons for unfavorable treatment outcome is that LLMD are often accompanied with cognitive impairment (attention, processing speed, memory and executive function) during an episode and after remission.This cognitive impairment in LLMD is associated with worse social functioning , distress to patients and caregivers, decreased quality of life and an unfavorable prognosis, including nursing home admission.

Several dimensions of recovery can be distinguished and are known to influence each other. For example, addressing functional recovery by improving cognitive functioning may enhance clinical recovery (less mood symptoms) and social functioning . Therefore, addressing cognitive impairment in LLMD may improve overall functioning and recovery rates.

Strategies to improve cognitive functioning with cognitive training and/or remediation are lacking for LLMD. Cognitive training has been effective in healthy older adults and in patients with mild cognitive impairment (MCI) and dementia.

A meta-analysis of adult patients with major depressive disorder showed that computerized cognitive training is associated with improvement in depressive symptoms and everyday functioning, though effects on cognition are inconsistent, with moderate to large effects for attention, working memory and global functioning and no effects for executive functioning and verbal memory. However, a small study including both unipolar and bipolar adult patients (n=15) and a control group (n=16) observed improvements in shifting, divided attention, global executive control after an online cognitive training. In addition, improved subjective cognitive functioning, reduced depression levels and less difficulty in everyday coping were observed.

In sum, cognitive impairment is a core feature of LLMD, contributes markedly to disability but is overlooked in current evidence-based treatment programs and therefore a less positive prognosis for these patients. An effective evidence-based treatment approach addressing cognitive impairment in LLMD is warranted.

AIM To age successfully, effective coping styles and social and community involvement are important. In the general population social activities and memory training are promoted for older persons as strategies to optimize resilience and to prolong independent living. Nevertheless, for the increasing number of patients with LLMD, effective interventions to improve cognition and social functioning are not available.

With the proposed pilot study we aim to seek a feasible and effective treatment to improve cognition, social functioning and quality of life of our patients. We aim to evaluate the feasibility of the online cognitive training (BrainGymmer) in a double-blind randomized control pilot-study.

If proven to be feasible, our intention is to expand the current pilot study to a RCT to test the efficacy of the proposed online cognitive training in patients with LLMD. After efficacy has been proven, the cognitive training program can also be used in other mental health departments, and even be made available through initiatives such as GGD appstore and onlinehulpstempel.nl.

OUTCOME At baseline, after the intervention period and 3 months after training, measurements will be taken. Our primary outcome measures will feasibility and appreciation of the intervention. Evaluation of therapy compliance, drop-out, and evaluation of the patients will be done with use of questionnaires on difficulty, feasibility, joy, effort, challenge of the therapy and clearness of the intervention explanation. Furthermore, evaluation groups (also mirror groups) will be held. In these discussion groups we will evaluate the study together with patients.

Secondary outcome measures include subjective and objective cognitive functioning, mood symptoms social functioning, quality of life and sense of Mastery.

ELIGIBILITY:
Inclusion Criteria:

* 50 years and older
* subjective cognitive complaints
* early or partial remission of depressive episode with a diagnosis of unipolar recurrent depression (current episode is at least the third episode and shorter than 2 years) or bipolar disorder according to DSM 5 criteria.
* have acces to internet on computer, tablet or lapyop
* willing to sign informed consent

Exclusion Criteria:

* current psychotic symptoms
* severe suicidal ideations
* severe personality disorder (as a main diagnosis)
* severe alcohol or substance abuse
* insufficient mastery of the Dutch language.
* on 2 or more cognitive domains below 1 SD of the norm
* moca < 22

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2019-09-17 (Actual); Primary Completion 2021-11-11 (Actual); Study Completion 2021-11-11 (Actual)

PRIMARY OUTCOMES:
Feasability of the intervention measured via therapy compliance and drop-out | Eight weeks (T1)
  therapy compliance, drop-out
Appreciation of the intervention | Eight weeks (T1)
  Questionnaire on difficulty, feasability, joy, effort, challenge of the therapy, clearness of the intervention explanation, evaluation groups (mirror groups)

SECONDARY OUTCOMES:
Subjective cognitive functioning measured via the CFQ | Eight weeks (T1) and 3 months (T2)
  Cognitive failures Questionnaire
Genaral objective cognitive functioning via the MOCA | Eight weeks (T1) and 3 months (T2)
  Montreal Cognitive Assessment
Mood symptoms via MADRS | Eight weeks (T1) and 3 months (T2)
  Montgomery Asberg Depression Rating Scale
Quality of life via the MANSA | Eight weeks (T1) and 3 months (T2)
  Manchester Short Assessment of quality of Life
Sense of Mastery via Mastery questionnaire | Eight weeks (T1) and 3 months (T2)
  Mastery questionnaire
Physical activity via NZPAQ-SF | Eight weeks (T1) and 3 months (T2)
  New Zealand Physical Activity Questionnaire - Short Form
Believe and expectancy of the intervention via credibility/expectancy questionnaire | Week 0 (T0)
  credibility/expectancy questionnaire
Social andf occupational functioning via SOFAS | Eight weeks (T1) and 3 months (T2)
  social and occupation functioning assessment scale

OTHER OUTCOMES:
Apathy via apathy scale | Eight weeks (T1) and 3 months (T2)
  apathy scale
Global cognitive dysfunction via the Pentagon Drawing Test | Eight weeks (T1) and 3 months (T2)
  Pentagon Drawing Test
Information processing speed and inhibition via the STROOP-test | Eight weeks (T1) and 3 months (T2)
  STROOP-test
Verbal functioning via verbal letter fluency test | Eight weeks (T1) and 3 months (T2)
  verbal letter fluency test
Cognitive functioning via SDMT | Eight weeks (T1) and 3 months (T2)
  symbol digit modalitities test
Cognitive functioning via VAT | Eight weeks (T1) and 3 months (T2)
  Verbal Assessment Test
Cognitive functioning via TMT | Eight weeks (T1) and 3 months (T2)
  trail making test
Cognitive functioning via 15-Woordentest | Eight weeks (T1) and 3 months (T2)
  15-Woordentest
Cognitive functioning via BNT short version - 30 | Eight weeks (T1) and 3 months (T2)
  Boston naming test, short version
Cogntive functioning via category fluency test | Eight weeks (T1) and 3 months (T2)
  category fluency test

CONTACTS AND LOCATIONS:
Overall Officials: Annemiek Dols, MD, PhD, Principal Investigator — Amsterdam UMC, location VUmc; Mardien Oudega, MD, PhD, Principal Investigator — Amsterdam UMC, location VUmc
Locations (1):
- GGZ inGeest, Amsterdam, North Holland, Netherlands

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Depp C, Vahia IV, Jeste D. Successful aging: focus on cognitive and emotional health. Annu Rev Clin Psychol. 2010;6:527-50. doi: 10.1146/annurev.clinpsy.121208.131449. PMID 20192798
- [Background] Farrand P, Matthews J, Dickens C, Anderson M, Woodford J. Psychological interventions to improve psychological well-being in people with dementia or mild cognitive impairment: systematic review and meta-analysis protocol. BMJ Open. 2016 Jan 27;6(1):e009713. doi: 10.1136/bmjopen-2015-009713. PMID 26817638
- [Background] Harris Y, Cooper JK. Depressive symptoms in older people predict nursing home admission. J Am Geriatr Soc. 2006 Apr;54(4):593-7. doi: 10.1111/j.1532-5415.2006.00687.x. PMID 16686868
- [Background] Korten NC, Penninx BW, Kok RM, Stek ML, Oude Voshaar RC, Deeg DJ, Comijs HC. Heterogeneity of late-life depression: relationship with cognitive functioning. Int Psychogeriatr. 2014 Jun;26(6):953-63. doi: 10.1017/S1041610214000155. Epub 2014 Feb 24. PMID 24565278
- [Background] Kuiper JS, Zuidersma M, Zuidema SU, Burgerhof JG, Stolk RP, Oude Voshaar RC, Smidt N. Social relationships and cognitive decline: a systematic review and meta-analysis of longitudinal cohort studies. Int J Epidemiol. 2016 Aug;45(4):1169-1206. doi: 10.1093/ije/dyw089. Epub 2016 Jun 6. PMID 27272181
- [Background] Motter JN, Pimontel MA, Rindskopf D, Devanand DP, Doraiswamy PM, Sneed JR. Computerized cognitive training and functional recovery in major depressive disorder: A meta-analysis. J Affect Disord. 2016 Jan 1;189:184-91. doi: 10.1016/j.jad.2015.09.022. Epub 2015 Sep 26. PMID 26437233
- [Background] Preiss M, Shatil E, Cermakova R, Cimermanova D, Ram I. Personalized cognitive training in unipolar and bipolar disorder: a study of cognitive functioning. Front Hum Neurosci. 2013 May 13;7:108. doi: 10.3389/fnhum.2013.00108. eCollection 2013. PMID 23717272
- [Background] Radua J, Grunze H, Amann BL. Meta-Analysis of the Risk of Subsequent Mood Episodes in Bipolar Disorder. Psychother Psychosom. 2017;86(2):90-98. doi: 10.1159/000449417. Epub 2017 Feb 10. PMID 28183076
- [Background] Schouws SN, Stek ML, Comijs HC, Dols A, Beekman AT. Cognitive decline in elderly bipolar disorder patients: a follow-up study. Bipolar Disord. 2012 Nov;14(7):749-55. doi: 10.1111/bdi.12000. Epub 2012 Sep 21. PMID 22998105
- [Background] Spijker, J., Bockting, C.L.H., Meeuwissen, J.A.C., et al. (2013) Dutch Multidisciplinary guideline for Depression: Trimbos Institute.
- [Background] Strohle A, Schmidt DK, Schultz F, Fricke N, Staden T, Hellweg R, Priller J, Rapp MA, Rieckmann N. Drug and Exercise Treatment of Alzheimer Disease and Mild Cognitive Impairment: A Systematic Review and Meta-Analysis of Effects on Cognition in Randomized Controlled Trials. Am J Geriatr Psychiatry. 2015 Dec;23(12):1234-1249. doi: 10.1016/j.jagp.2015.07.007. Epub 2015 Jul 21. PMID 26601726
- [Background] van der Stel JC. [Functional recovery and self-regulation: assignments for both clients and psychiatrists]. Tijdschr Psychiatr. 2015;57(11):815-22. Dutch. PMID 26552928
- [Background] van Liempt S, Dols A, Schouws S, Stek ML, Meesters PD. Comparison of social functioning in community-living older individuals with schizophrenia and bipolar disorder: a catchment area-based study. Int J Geriatr Psychiatry. 2017 May;32(5):532-538. doi: 10.1002/gps.4490. Epub 2016 Apr 27. PMID 27121916
- [Background] Willis SL, Tennstedt SL, Marsiske M, Ball K, Elias J, Koepke KM, Morris JN, Rebok GW, Unverzagt FW, Stoddard AM, Wright E; ACTIVE Study Group. Long-term effects of cognitive training on everyday functional outcomes in older adults. JAMA. 2006 Dec 20;296(23):2805-14. doi: 10.1001/jama.296.23.2805. PMID 17179457
- [Background] Yliruka, L. (2012) 'The Mirror Method: a structure supporting expertise in social welfare services.', Social Work & Social Sciences Review., 15(2), pp. 9-37.
- [Derived] Oudega ML, Wagenmakers MJ, Palsma T, Hoogendoorn AW, Vriend C, van den Heuvel OA, Schouws S, Dols A. BrainFit: improving executive and subjective cognitive functioning in late-life mood disorders - a double-blind randomized active-controlled study evaluating the effect of online cognitive training. Front Psychiatry. 2025 Jan 2;15:1509821. doi: 10.3389/fpsyt.2024.1509821. eCollection 2024. PMID 39822386